CLINICAL TRIAL: NCT05758558
Title: Cognitive, Psychological, and Physical Functioning in Long-COVID Patients With Different Levels of Fatigue.
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Stef Feijen, Doctoral Assistant, Hasselt University
Other Study IDs: CME2022/021 S66200
Record Dates: First submitted 2023-02-08; First posted 2023-03-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post COVID-19 usually occurs 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Patients report a range of disabling symptoms such as fatigue, shortness of breath, cognitive impairment, memory loss and mental health and employment issues. This clinical heterogeneity complicates the identification of the appropriate needs and care.

The aim of this cross-sectional study is to identify subgroups (clusters) of post COVID patients based on clinical symptoms, demographic characteristics, levels of fatigue and physical, cognitive and psychological functioning of the individuals.

ELIGIBILITY:
Inclusion Criteria:

The participant must report current persisting symptoms (such as brain fog, anxiety, shortness of breath, headaches but also others) and indicate on the Post COVID-19 Functional Status Scale that these have an impact on everyday functioning (grade 2, 3, and 4). These symptoms need to be present for more than two months.

Further inclusion criteria are:

* Fatigue Severity Scale (FSS) score > 4
* Aged over 18 years old
* Willing to sign the digital informed consent
* Dutch speaking and Dutch understanding
* Be tested positive for COVID-19, i.e. by reverse transcription polymerase chain reaction (RT-PCR), computed tomography (CT) of the lungs, or symptom-based diagnosis by the general practitioner.

Exclusion Criteria:

* Pregnant women
* Pacemaker, defibrillator
* Brain or nerve disorders
* Epilepsy
* A copper spiral or recent bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that match the criteria of the recently published definition of the post-COVID-19 condition will be considered eligible to participate in the study.[8] Post-COVID-19 has been defined as a condition that occurs in individuals with a history of confirmed SARS-CoV-2 infection, and that occurs usually within three months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis. Consequently, participants that either have or have not been hospitalized will both be allowed to participate in this study. COVID infection will be self-reported by the participant. Participants will be encouraged to show any test certificate but they are not obligated to do so.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Physical evaluation | Day 1
  Hand grip strength (Jamar hand dynamometer) & Six Minute Walk Test (6MWT)
Fatigue severity | Day 1
  Fatigue severity scale (FSS)
Psychological evaluation | Day 1
  Anxiety and depression Scale (HADS); MINI-S, MINI International Neuropsychiatric Interview - Simplified (Overbeek & Schruers 2019)
Cognitive evaluation | Day 1
  Multi-modal Evaluation of Sensory Sensitivity (MESSY); Montreal Cognitive Assessment (MoCA)

OTHER OUTCOMES:
Number of clusters | Day 1
  The main outcome of the study is identification of the best-fitting number of clusters and the reliability of clustering. To check for differences in characteristics between the clusters, we will use an analysis of variance for normally distributed continuous variables and the nonparametric Kruskal-Wallis test for nonnormally variances (R package "FSA").

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: Undecided